CLINICAL TRIAL: NCT02137018
Title: "Nanotechnologies Applied to General Surgery and Emergency Surgery: The Buckypaper as a New Fixing Method for Prosthetic Materials in the Treatment of Abdominal Wall Hernias, Diaphragmatic Hernias, Diaphragmatic Rupture, Incisional Hernia and Abdominal Wall Disaster in Laparotomy Procedure and Laparoscopic Procedures".
Brief Title: "Nanotechnologies Applied to General Surgery and Emergency Surgery: Buckypaper as a New Fixing Method for Prosthetic Materials for the Treatment of Hernia and Incisional Hernia in Laparotomy and Laparoscopic
Acronym: 36P
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Martinelli, Andrea, M.D. (Individual); GA Carru (Unknown); AM Chiaretti (Unknown); F Faiola (Unknown); G Ceccarelli (Unknown); AI Chiaretti (Unknown); P Consentino (Unknown); E Valente (Unknown)
Responsible Party: Principal Investigator, Massimo Chiaretti, Researcher, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36Pa
Record Dates: First submitted 2014-05-06; First posted 2014-05-13 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2014-05

CONDITIONS: Hernia; Incisional Hernia
Keywords: hernia; incisional hernia; device; pig
MeSH Terms: conditions — Hernia; Incisional Hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- laparotomy with PPL mesh implantation (Active Comparator): control group: laparotomy with PPL mesh implantation (traditional method)
  Interventions: Device: PPL mesh
- laparotomy with PPL fixation by BP (Experimental): laparotomic surgery with PPL mesh fixation by BP (new fixing method)
  Interventions: Device: PPL fixation by BP
- laparoscopy with PPL mesh implantation (Active Comparator): control group: laparoscopy with PPL mesh implantation (traditional method)
  Interventions: Device: PPL mesh
- laparoscopy with PPL fixation by BP (Experimental): laparoscopic surgery with PPL mesh fixation by BP (new fixing method)
  Interventions: Device: PPL fixation by BP

INTERVENTIONS:
Device: PPL fixation by BP — A surgical scar was performed on the abdominal linea alba and carried out deeply into a pocket between large abdominal muscle and abdominal fascia. A pocket was created between the two layers. 5cm PLL prosthesis was implanted and fixed by BP patch. The scar was sutured with absorbable stitches on subcutaneous incision and not absorbable stitches on the cutaneous layer.
  Other Names: PPL Premilene mesh B Braun (ref. 1064435, lot. 112313); PPL Parietene mesh Tyco (ref. PP3030, lot. SIK00587); V-Loc 180 (ref. VLOCL0024, lot. A1D0998); The BP (NanoLab Inc, Newton, MA 02458 USA)
  Arms: laparoscopy with PPL fixation by BP; laparotomy with PPL fixation by BP
Device: PPL mesh — A surgical scar was performed on the abdominal linea alba and carried out deeply into a pocket between large abdominal muscle and abdominal fascia. A pocket was created between the two layers. 5cm PLL prosthesis was implanted and fixed by absorbable stichtes. The scar was sutured with absorbable stitches on subcutaneous incision and not absorbable suture on the cutaneous layer.
  Other Names: PPL Premilene mesh B Braun (ref. 1064435, lot. 112313); PPL Parietene mesh Tyco (ref. PP3030, lot. SIK00587); V-Loc 180 (ref. VLOCL0024, lot. A1D0998)
  Arms: laparoscopy with PPL mesh implantation; laparotomy with PPL mesh implantation

SUMMARY:
"Nanotechnologies applied to General Surgery and Emergency Surgery: The Buckypaper as a new fixing method for prosthetic materials in the treatment of abdominal wall hernias, diaphragmatic hernias, diaphragmatic rupture, incisional hernia and abdominal wall disaster in laparotomy procedure and laparoscopic procedures". Experimentation on breed pig Lantrace ANIMAL MODEL.

ELIGIBILITY:
Inclusion Criteria:

* animal model: lantrace female pigs of 20 kg of body weight

Exclusion Criteria:

* any kind of illness in porcine subjects

Ages: 3 Months to 6 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Time of durability without side effects of surgical device | up to 36 months
  We are testing the time (months/year) of durability without side effects of a new fixing method for prosthetic materials for abdominal wall hernias and wall defects repairing on pig model

SECONDARY OUTCOMES:
time required to position the device during surgery | up to 36 months
  time required to position the device during surgery (time is related with probability of side effect during surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Chiaretti, MD, PhD, MSc, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Animal House Agostino Gemelli University of Rome., Rome, RM, Italy

REFERENCES:
- [Background] Martinelli A, Carru GA, D'Ilario L, Caprioli F, Chiaretti M, Crisante F, Francolini I, Piozzi A. Wet adhesion of buckypaper produced from oxidized multiwalled carbon nanotubes on soft animal tissue. ACS Appl Mater Interfaces. 2013 May 22;5(10):4340-9. doi: 10.1021/am400543s. Epub 2013 May 1. PMID 23635074
- [Background] Bellucci S, Chiaretti M, Onorato P, Rossella F, Grandi MS, Galinetto P, Sacco I, Micciulla F. Micro-Raman study of the role of sterilization on carbon nanotubes for biomedical applications. Nanomedicine (Lond). 2010 Feb;5(2):209-15. doi: 10.2217/nnm.09.100. PMID 20148633
- [Background] Bellucci S, Chiaretti M, Cucina A, Carru GA, Chiaretti AI. Multiwalled carbon nanotube buckypaper: toxicology and biological effects in vitro and in vivo. Nanomedicine (Lond). 2009 Jul;4(5):531-40. doi: 10.2217/nnm.09.36. PMID 19572819
- [Background] Di Sotto A, Chiaretti M, Carru GA, Bellucci S, Mazzanti G. Multi-walled carbon nanotubes: Lack of mutagenic activity in the bacterial reverse mutation assay. Toxicol Lett. 2009 Feb 10;184(3):192-7. doi: 10.1016/j.toxlet.2008.11.007. Epub 2008 Nov 21. PMID 19063954